CLINICAL TRIAL: NCT07394985
Title: Fiability of a Telerehabilitation Programme Based on the Neurodevelopmental Treatment (NDT) Model on Gross Motor Function and Functional Performance in Children With Cerebral Palsy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior Saúde Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Olga Maria Barros Maia, Olga Maria Barros Maia, Escola Superior Saúde Fernando Pessoa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESTUDO_PC_TELEREAB_01
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy Children

STUDY DESIGN:
Intervention Model Description: This is a parallel-group experimental study in which participants are assigned to an intervention group or a control group. The intervention group undergoes a structured telerehabilitation program based on neurodevelopmental principles, while the control group continues with usual care. Outcome measures are collected at baseline and post-intervention to assess changes within each group over time.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): telerhabilitation intervention in accordance with neurodevelopmental treatment
  Interventions: Other: neurodevelopmental treatment based on the Bobath concept
- Control Group (Experimental): face-to-face intervention in accordance with neurodevelopmental treatment
  Interventions: Other: neurodevelopmental treatment according to the Bobath concept

INTERVENTIONS:
Other: neurodevelopmental treatment based on the Bobath concept — Participants in the intervention group receive a structured telerehabilitation program based on neurodevelopmental principles. The intervention is delivered remotely by a physiotherapist through scheduled sessions and focuses on improving motor control, postural alignment, balance, and functional movement according to each child's abilities. The program is individualized and adapted to the functional level of each participant and is conducted over a predefined intervention period.
  Arms: Intervention Group
Other: neurodevelopmental treatment according to the Bobath concept — Participants in the control group continue to receive conventional in-person physiotherapy based on neurodevelopment according to the Bobath concept.
  Arms: Control Group

SUMMARY:
Experimental study with a control group, developed with the aim of analyzing the impact of a telerehabilitation program based on the Neurodevelopmental Treatment (NDT) model on gross motor function and functional performance in children with cerebral palsy.

DETAILED DESCRIPTION:
The sample consisted of 20 children divided into two equivalent groups: an experimental group (n = 10), which received the TND intervention program in a synchronous telerehabilitation format for six months, and a control group (n = 10), which maintained the usual care and clinical follow-up plan without additional structured intervention.

The children included had a clinical diagnosis of spastic cerebral palsy, aged between 6 months and 6 years, classified between levels I and IV of the Gross Motor Function Classification System (GMFCS).

The pre-intervention assessment was performed before the start of the program, and the post-intervention assessment took place after six months. The assessments included the GMFM-88, to measure gross motor function, and the CO-OP Performance Measure (COOPM), to assess caregivers' perceptions of performance and satisfaction.

ELIGIBILITY:
Inclusion criteria Confirmed diagnosis of cerebral palsy; Age between 6 months and 6 years; Ability of the primary caregiver to actively participate in online sessions; Regular access to a device with a camera and internet connection.

Exclusion criteria Orthopaedic surgery or botulinum toxin application in the six months prior to the intervention; Presence of severe comorbidities (cardiorespiratory, cognitive, or sensory) that would limit participation;

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | Baseline and at the end of the 6-month intervention period
  instrument designed to evaluate changes in gross motor abilities in children with cerebral palsy.
Gross Motor Function Measure (GMFM-88) | Baseline and at the end of the 6-month intervention period
  Gross motor function assessed using the Gross Motor Function Measure-88 (GMFM-88), a validated observational instrument designed to evaluate changes in gross motor abilities in children with cerebral palsy.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Baseline and at the end of the 6-month intervention period
  Occupational performance and satisfaction assessed using the Canadian Occupational Performance Measure (COPM), administered to the child's primary caregiver as a proxy respondent. Caregivers identify meaningful daily activities and rate the child's performance and satisfaction on a 10-point scale. Changes from baseline to post-intervention are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Associação do Porto de Paralisia Cerebral, Porto, Porto District, Portugal